CLINICAL TRIAL: NCT04268979
Title: Electronic Social Network Assessment Program (eSNAP) + Caregiver Navigator Intervention for Neuro-Oncology
Brief Title: Electronic Social Network Assessment Program (eSNAP) + Caregiver Navigator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC 19731; 5R01CA236034-05 (NIH)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Brain Cancer
Keywords: Neuro Oncology
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eSNAP & Caregiver Navigator (Experimental): eSNAP intervention plus questionnaires
  Interventions: Behavioral: eSNAP; Behavioral: Caregiver Navigator
- Waitlist Control Condition (No Intervention): Participants randomly assigned to the waitlist control condition will only complete questionnaires during the 8-week study period. After the 8 weeks, they will then have access to the eSNAP, including completion of questionnaires and 8 weeks of Caregiver Navigator sessions as needed.

INTERVENTIONS:
Behavioral: eSNAP — eSNAP is a web based tool that quickly collects and organizes social support information entered by Family Caregivers (FCGs) into visualizations of the size, quality, and function of support networks. Visualizations can help FCGs catalogue support resources and present them in a new way, which may make them more salient and remind FCGs of their availability.
  Other Names: Electronic Social Network Assessment Program
  Arms: eSNAP & Caregiver Navigator
Behavioral: Caregiver Navigator — The Caregiver Navigator will have social work training and will help Family Caregivers (FCGs) identify and leverage informal and formal social support, including enrolling or directing FCGs to services.
  Arms: eSNAP & Caregiver Navigator

SUMMARY:
The purpose of the study is to determine if family caregivers of neuro-oncology patients feel less burdened by utilizing the Electronic Social Network Assessment Program (eSNAP) + the Caregiver Navigator.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking/reading/writing
* Able to complete questionnaires (including by proxy)
* Family Caregivers (FCGs) must self-identify as being a primary FCG of a patient with a primary brain tumor, secondary (metastatic) brain tumor, or leptomeningeal disease diagnosis. A primary caregiver is a family member, friend, or other unpaid person who provides at least some care for a patient at home.
* Patients must be diagnosed with new or recurrent primary brain tumor, a secondary (metastatic) brain tumor or leptomeningeal disease within the last 9 months, receiving at least some evaluation and/or care at Moffitt (i.e. at least one appointment), have a prognosis of at least 9 months

Exclusion Criteria:

* Patients may not participate without a consenting FCG, but FCGs may participate without a consenting patient
* Patients and FCGs who are experiencing acute distress will be excluded from enrollment and referred directly to social work, per Moffitt policy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Byrne, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- [Derived] Reblin M, Wells KJ, Zebrack BJ, Witte D, Byrne MM. Associations of Critical Relationships With Distress and Burden in Caregivers of Patients With Brain Tumor. Psychooncology. 2025 Nov;34(11):e70332. doi: 10.1002/pon.70332. PMID 41198147
- [Derived] Reblin M, Ketcher D, McCormick R, Barrios-Monroy V, Sutton SK, Zebrack B, Wells KJ, Sahebjam S, Forsyth P, Byrne MM. A randomized wait-list controlled trial of a social support intervention for caregivers of patients with primary malignant brain tumor. BMC Health Serv Res. 2021 Apr 17;21(1):360. doi: 10.1186/s12913-021-06372-w. PMID 33865382

RESULTS

PARTICIPANT FLOW:
Groups:
- Family Caregivers: Family caregivers (FCGs) of patients with a primary brain tumor, secondary (metastatic) brain tumor, or leptomeningeal disease.
- Neuro Patients: Patients diagnosed with a new or recurrent primary brain tumor, a secondary (metastatic) brain tumor, or leptomeningeal disease within the last 9 months, and receiving at least some evaluation and/or care at Moffitt.
Period: Overall Study
Arm/Group | Family Caregivers | Neuro Patients
Started | 148 | 148
Completed | 102 | 89
Not Completed | 46 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Family Caregivers | Neuro Patients | Total
Number analyzed (Participants) | 148 | 148 | 296
Age, Continuous [Mean (Full Range); unit: years] — Population: Only partial healthy care giver demographic data is available for baseline measures since they do not have a medical record
  years
    number analyzed (Participants) | 122 | 148 | 270
    (all) | 57.1 [23 to 85] | 58.2 [22 to 87] | 57.7 [22 to 87]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only partial healthy care giver demographic data is available for baseline measures since they do not have a medical record
  Participants
    number analyzed (Participants) | 124 | 148 | 272
    Female | 87 | 68 | 155
    Male | 37 | 80 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 113 | 131 | 244
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 26 | 9 | 35
Region of Enrollment [Number; unit: participants]
  United States | 148 | 148 | 296

OUTCOME MEASURES:

1. Primary Outcome: Family Caregiver Well-Being Using GAD-7 Scale
Description: Caregiver well being will be measured using the Generalized Anxiety Disorder 7 Item Scale (GAD-7). The GAD-7 measures anxiety scoring 0-3 points per item, with a total score range 0-21,with a higher score meaning more anxiety.
Time Frame: 8 weeks per participant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers
Number analyzed (Participants) | 94
score on a scale | 8.95 (6.08)

2. Primary Outcome: Family Caregiver Well-Being Using PHQ-8 Scale
Description: Caregiver well being will be measured using the Personal Health Questionnaire Depression 8 Item Scale Scale (PHQ 8). The PHQ 8 measures depression scoring 0-3 points per item, with a total score range of 0-24, with the higher score meaning more depression.
Time Frame: 8 weeks per participant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers
Number analyzed (Participants) | 94
score on a scale | 7.11 (5.45)

3. Primary Outcome: Family Caregiver Well-Being Using Zarit Burden Interview
Description: Caregiver well being will be measured using the Zarit Burden Interview. The Zarit Burden Interview measures burden scoring 0-4 points per item, with a total score range of 0-48, with the higher score meaning more burden.
Time Frame: 8 weeks per participant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers
Number analyzed (Participants) | 94
score on a scale | 13.77 (9.15)

4. Primary Outcome: Neuro Patients Well-Being Using GAD-7 Scale
Description: Neuro patients well being will be measured using the Generalized Anxiety Disorder 7 Item Scale (GAD-7). The GAD-7 measures anxiety scoring 0-3 points per item, with a total score range 0-21,with a higher score meaning more anxiety.
Time Frame: 8 weeks per participant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuro Patients
Number analyzed (Participants) | 56
score on a scale | 5.66 (5.40)

5. Primary Outcome: Neuro Patients Well-Being Using PHQ-8 Scale
Description: Neuro patients well being will be measured using the Personal Health Questionnaire Depression 8 Item Scale Scale (PHQ 8). The PHQ 8 measures depression scoring 0-3 points per item, with a total score range of 0-24, with the higher score meaning more depression.
Time Frame: 8 weeks per participant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neuro Patients
Number analyzed (Participants) | 56
score on a scale | 7.91 (5.77)

6. Primary Outcome: Neuro Patients Well-Being Using NeuroQol
Description: Neuro patients well being will be measured using Neuro-Qol (Neuro Quality of Life) which will be using T scores where the lower values represent worse outcomes. 50 indicates the population mean with a standard deviation of 10.
Time Frame: 8 weeks per participant
Measure: Mean (Standard Error); unit: T-Score
Arm/Group | Neuro Patients
Number analyzed (Participants) | 86
T-Score | 40.9 (2.6)

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Family Caregivers | Neuro Patients
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT04268979/Prot_SAP_000.pdf